CLINICAL TRIAL: NCT01668862
Title: A Prospective, Multicentric, Open Label, Randomised, Bio-Interventional Phase I/II Pilot Study To Evaluate The Safety And Efficacy Of Autologous Human Platelet Lysate (HPL) For The Treatment Of Lateral Epicondylitis (Tennis Elbow)
Brief Title: A Study to Determine Safety & Efficacy of Autologous Human Platelet Lysate in Lateral Epicondylitis (Tennis Elbow)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasiak Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRPL/HPL-TE/11-12/003
Record Dates: First submitted 2012-07-17; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-07

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
MeSH Terms: conditions — Tennis Elbow | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study arm A (Other): Subjects will receive one injection of Autologous Human Platelet lysate in the lateral epicondyle space
  Interventions: Biological: Autologous Human Platelet Lysate
- Control Arm B (Other): Subjects will receive one injection of Corticosteroid in the lateral epicondyle space
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Biological: Autologous Human Platelet Lysate — Subjects will receive one injection of Autologous Human Platelet Lysate in the lateral epicondyle space
  Arms: Study arm A
Drug: Corticosteroid — Subjects will receive one injection of Corticosteroid in the lateral epicondyle space
  Arms: Control Arm B

SUMMARY:
This is a multicentre, open label, randomized, pilot study to evaluate safety and efficacy of human Platelet Lysate (HPL) in subjects with Lateral Epicondylitis (Tennis Elbow). The study is being conducted in 2 centers in India. The primary end points are Visual Analog Score (VAS) and Patient rated tennis elbow evaluation (PRTEE) score. The secondary endpoint is improvement in ultrasonography form randomization to End of study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinical diagnosis of tennis elbow within the last 3 months
* Subjects both male and female, aged 18-60 years (both inclusive)
* Subjects who are willing to give informed consent and adhere to the study protocol

Exclusion Criteria:

* Subjects aged less than 18 and more than 60 years
* Subjects with autoimmune diseases
* Subjects with immuno-compromised system
* Subjects on Anti-coagulant therapy or blood thinning medicines like Aspirin
* Subjects taking concomitant therapy that might interfere with the study results in investigators opinion or who had concomitant other injury of the tennis elbow tendons.
* Subjects who have received treatment with corticosteroid injections within the last 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Score (VAS) | Day 0, Month 1, Month 2, End of Study - Month 3

SECONDARY OUTCOMES:
Change in Ultrasonography of the lateral epicondyle region from Baseline to End of study at Month 3 | Day 0, End of study - Month 3

OTHER OUTCOMES:
Patient rated tennis elbow evaluation (PRTEE Score) | Day 0, Month 1, Month 2, End of study-Month 3
The American Shoulder and Elbow Society score | Dya 0, Month 1, Month 2, End of study-Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Anant Joshi, Dr., Principal Investigator — ASMI; Nicolas Antao, Dr., Principal Investigator — Hillway Clinic; Gauresh Palekar, Dr., Principal Investigator — Surya Orthopedic Clinic
Locations (1):
- Kasiak Research Pvt Ltd, Thane, Maharashtra, India